CLINICAL TRIAL: NCT04247477
Title: Comparison of Different Positive End-expiratory Pressure Titration Strategies Using ELectrical Impedance Tomography in Patients With Acute Respiratory Distress Syndrome : the DELTA Physiological Study
Brief Title: Comparison of Different PEEP Titration Strategies Using Electrical Impedance Tomography in Patients With ARDS
Acronym: DELTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 49RC19_0249
Record Dates: First submitted 2020-01-21; First posted 2020-01-30 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome); Electrical Impedance Tomography (EIT); Positive End Expiratory Pressure (PEEP); Acute Lung Injury
Keywords: ARDS; EIT; PEEP titration; Mechanical Ventilation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Intervention Model Description: We use a crossover sequential model, with all 3 strategies tested in both arms.
  A reference strategy, based on the Express method (PEEP level adjusted to reach a plateau pressure of 28-30 cmH2O), is applied at the begining of the study and during a wash-out period (between the 2 periods of application of the 2 EIT-based strategies).
  The 2 EIT-based strategies are applied in a randomized order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-B-A-C (Experimental): Four consecutive steps (45 min per step) are tested in the following order: Peep titration strategy according to Express method (A) - Peep titration strategy according to overdistension and collapse estimation (B) - Peep titration strategy according to Express method (A) - Peep titration strategy according to estimation of lung inhomogeneity (C)
  Interventions: Other: Ventilation strategy
- A-C-A-B (Experimental): Four consecutive steps (45 min per step) are tested in the following order: Peep titration strategy according to Express method (A) - Peep titration strategy according to estimation of lung inhomogeneity (C) - Peep titration strategy according to Express method (A) - Peep titration strategy according to overdistension and collapse estimation (B)
  Interventions: Other: Ventilation strategy

INTERVENTIONS:
Other: Ventilation strategy — Patients are ventilated in randomized order with three different ventilation strategies (A,B and C)

SUMMARY:
The aim of the this study is to assess the short term physiological effects of 3 ventilation strategies for adult patients with ARDS admitted to intensive care unit.

Two of those strategies are based on electrical impedance tomography (EIT) monitoring.

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate to severe ARDS, defined by the Berlin consensus, at 12 to 48h from diagnosis
* PaO2/FiO2 ratio < 150 mmHg
* Patient affiliated to or beneficiary of a health care plan
* Consent obtained from patient's SDM

Exclusion Criteria:

* Pneumothorax
* Contraindication to the insertion of a nasogastric tube with an esophageal balloon
* Contraindication to the use of Electrical impedance tomography
* Pregnancy, lactating or parturient woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Change in PaO2 (mmHg) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance!

SECONDARY OUTCOMES:
Change in PaCO2 (mmHg) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Plateau pressure (cmH2O) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Positive end expiratory pressure (cmH2O) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Expiratory and inspiratory transpulmonary pressure (cmH2O) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Regional ventilation distribution (%) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Center of ventilation (%) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Overdistension and collapsus (%) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Global and regional end expiratory lung impedance changes (IU) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
End expiratory lung volume (mL) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Blood pressure (mmHg) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Heart rate (bpm) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance
Cardiac output (L/min) | Time : 0 ; 45 minutes ; 90 minutes ; 135 minutes ; 180 minutes
  As it is a physiological study, all the outcomes will be analyzed with the same importance

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France